CLINICAL TRIAL: NCT02951078
Title: A Study of Comparing Effects of Thulium Laser en Bloc Resection and Electrical Transurethral Resection of the Non-muscle Invasive Bladder Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Liu Haitao, Chief physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChiCTR-INR-16009513
Record Dates: First submitted 2016-10-23; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Thulium Laser en Bloc Resection of bladder tumor (Experimental): Thulium Laser en Bloc Resection of the Non-muscle Invasive Bladder tumor with thulium laser
  Interventions: Procedure: Thulium Laser en Bloc Resection of bladder tumor
- Electrical transurethral resection of bladder tumor (Active Comparator): Electrical transurethral resection of the Non-muscle Invasive Bladder tumor
  Interventions: Procedure: Electrical transurethral resection of bladder tumor

INTERVENTIONS:
Procedure: Thulium Laser en Bloc Resection of bladder tumor
  Arms: Thulium Laser en Bloc Resection of bladder tumor
Procedure: Electrical transurethral resection of bladder tumor
  Arms: Electrical transurethral resection of bladder tumor

SUMMARY:
This study is to verify the short-term efficacy and long-term prognosis of thulium laser resection compared with conventional transurethral resection of non-muscular invasive bladder cancer. Half of participants will receive thulium laser resection of bladder cancer, while the other half will receive electrical transurethral resection of bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological or histological diagnosis of primary non-muscle invasive bladder urothelial carcinoma (TaTisT1);
2. Imaging examinations showed the bladder muscle has not been affected, no lymph node metastasis or distant metastasis;
3. Patients who agree to TURBT surgery, and will be effected to the postoperative follow-up treatment such as conventional infusion after the operation;
4. Function of main organs (heart, liver, lung, kidney) should be normal, PS score 0-2;
5. Bladder capacity≥ 200ml.

Exclusion Criteria:

1. Find distant metastasis ,infiltration of the surrounding organs or relapse before operation.Metastatic bladder cancer or other cancers involve the bladder;
2. Received chemotherapy or BCG perfusion therapy in the nearly 3 months;
3. Patients who can not tolerate the serious side effects during the bladder perfusion treatment process (bladder irritation and other symptoms);
4. Patients during pregnancy ,critical care patients and patients who have other cases of surgical contraindications.Such as serious cardiovascular disease,coagulation abnormalities,non-transitional epithelial tumors( such as adenocarcinoma and squamous cell carcinoma),acute cystitis,can not be supine because of spinal deformity,untreated urethral stricture.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The residual rate of tumor in the second operation of the two surgical methods | 2 years